CLINICAL TRIAL: NCT03634709
Title: A Randomised Controlled Trial of Autobiographical Memory Flexibility Training (MemFlex) for Posttraumatic Stress Disorder
Brief Title: Autobiographical Memory Flexibility Training (MemFlex) for Posttraumatic Stress Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical Research Council Cognition and Brain Sciences Unit (Other Government)
Collaborators: Institute for Cognitive Science Studies, Iran (Unknown); Kharazmi University (Other)
Responsible Party: Principal Investigator, Caitlin Hitchcock, Senior Scientist, Medical Research Council Cognition and Brain Sciences Unit
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MemFlex for PTSD
Record Dates: First submitted 2018-02-23; First posted 2018-08-16 (Actual); Last update posted 2020-06-17 (Actual); Status verified 2020-04

CONDITIONS: Post Traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Single blind, randomized controlled trial comparing active intervention to waitlist control
Who Masked: Outcomes Assessor
Masking Description: Assessors will be blind to allocated condition
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Memory Flexibility Training (MemFlex) (Experimental): The MemFlex programme has been adapted from the initial format addressing depression-related memory distortions to facilitate completion with individuals experiencing posttraumatic stress. The workbook and associated materials have also been translated from English to Farsi. The programme consists of one researcher-facilitated session and eight self-guided workbook-based sessions that train memory retrieval skills and are completed over a one month period.
  Interventions: Behavioral: Memory Flexibility training (MemFlex)
- Waitlist control (No Intervention): After randomisation, the waitlist control group will be informed that they have been placed on a waiting list for the intervention. The participants will complete the baseline assessment and receive no further contact from the researcher until the post assessment one month later, followed by the follow-up assessment three months later. After the three month assessment, wait listed participants will receive the intervention. No further assessments will be completed.

INTERVENTIONS:
Behavioral: Memory Flexibility training (MemFlex) — MemFlex is a primarily self-guided, paper workbook-based program which aims to reduce overgeneral memory bias and improve recall of positive, specific event memories. Prior to completing one month of self-guided, workbook-based intervention, the participant will attend one 45 minute face-to-face session in which the facilitator outlines the importance of autobiographical memory in everyday life, discusses the impact of trauma on autobiographical memory, and provides information on the different types of autobiographical memories (e.g., specific, general) and their potential everyday functions. The session also introduces the cued-recall tasks which were used to train the memory skills throughout the workbook, and provides facilitator-assisted practice with the tasks. Once participants are comfortable with the training exercises, they set a schedule for completion of the eight-session workbook over the following four weeks.
  Arms: Memory Flexibility Training (MemFlex)

SUMMARY:
The experience of trauma not only impacts the way an individual thinks and feels, but can also produce changes in the way someone remembers their personal past. It is not only memories of the trauma that are affected- avoidance of trauma memories can also lead to memories of other events becoming vague, and in particular, memories of positive experiences can seem out of reach. This memory difficulty promotes posttraumatic stress disorder (PTSD). This study will explore an intervention that aims to improve memory difficulties, which should then flow on to improve PTSD. The study will be completed with individuals who have experienced a single incident trauma. Twenty five participants will complete MemFlex straight away, and 25 will go on a waiting list. Once this first group has finished MemFlex, the researchers will compare the two groups to see if the programme produced a larger reduction in PTSD symptoms. MemFlex is workbook-based, and as such, if it is successful it may offer an easy, cheap, and accessible way to offer psychological treatment to PTSD sufferers around the world.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Posttraumatic Stress Disorder (as indexed by the Farsi version of the Structured Clinical Interview for DSM disorders [SCID])
* Aged over 18 years

Exclusion Criteria:

* Lack of oral and/or written fluency in Farsi
* Traumatic brain injury or cognitive impairment, indexed via self-report
* Current experience of psychosis, indexed by SCID

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-08-19 (Actual); Primary Completion 2020-02-11 (Actual); Study Completion 2020-05-11 (Actual)

PRIMARY OUTCOMES:
Autobiographical memory | At post-intervention assessment (approximately 4-5 weeks after pre-intervention assessment)
  Number of correct responses on the Alternating Instructions Autobiographical Memory Test- Farsi version

SECONDARY OUTCOMES:
PTSD symptoms at post-intervention | At post-intervention assessment (approximately 4-5 weeks after pre-intervention assessment)
  Total score (range - 0-80) on the Farsi version of the Posttraumatic Stress Disorder Checklist for the Diagnostic and Statistical Manual of Mental Disorders- Fifth Edition
PTSD symptoms at follow-up | Three months following the completion of the intervention
  Total score (range - 0-80) on the Farsi version of the Posttraumatic Stress Disorder Checklist for the Diagnostic and Statistical Manual of Mental Disorders- Fifth Edition

OTHER OUTCOMES:
Posttraumatic Cognitions | At post-intervention assessment (approximately 4-5 weeks after pre-intervention assessment)
  Total score (range = 33-231) on the Farsi version of the Posttraumatic Cognitions Inventory
Trauma memory quality | At post-intervention assessment (approximately 4-5 weeks after pre-intervention assessment)
  Total score (range = 14-56) on the Farsi version of the Trauma Memory Quality Questionnaire
Rumination | At post-intervention assessment (approximately 4-5 weeks after pre-intervention assessment)
  Total score (range = 22-88) on the Farsi version of the Ruminative Response Scale
Depression | At post-intervention assessment (approximately 4-5 weeks after pre-intervention assessment)
  Total score (range = 0-63) on the Farsi version of the Beck Depression Inventory II
Future Thinking | At post-intervention assessment (approximately 4-5 weeks after pre-intervention assessment)
  Number of generated positive items on the Farsi version of the Future Thinking Task

CONTACTS AND LOCATIONS:
Locations (1):
- Institute for Cognitive Science Studies, Tehran, Iran

IPD SHARING:
Plan to Share IPD: Yes
De-identified dataset will be made available online and linked to the published results
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: At time of publication of peer-reviewed manuscript
Access Criteria: Open access